CLINICAL TRIAL: NCT05413343
Title: Clinical Study on Monitoring the Plasma Concentration of Ceftazidime-Avibactam in Critically Ill Patients
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-468
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-06

CONDITIONS: Severe Sepsis
Keywords: Severe sepsis; Ceftazidime-avibactam; Plasma drug concentration; Population pharmacokinetics (PPK); Pharmacokinetic (PK); Critically ill Patients; Pharmacodynamic (PD)
MeSH Terms: conditions — Sepsis | interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ceftazidime-avibactam — Patients with severe sepsis and treatment with CAZ-AVI will be enrolled. Blood samples at 0 hour, 2 hours, 4 hours, 6 hours, and 8 hours after the first time and the steady state concentration(more than 4 times drug administration) of drug administration will be collected to detect plasma drug concentrations of CAZ-AVI

SUMMARY:
A observational study is conducting at the First Affiliated Hospital of the Medical College of Zhejiang University from June 1, 2021 to January 1, 2024. Patients with severe sepsis and treatment with Ceftazidime-avibactam (CAZ-AVI) will be enrolled.

Blood samples at different time points: 0 hour, 2 hours, 4 hours, 6 hours, and 8 hours after the first time and the steady state concentration(more than 4 times drug administration) of drug administration will be collected to detect plasma drug concentrations of CAZ-AVI.

DETAILED DESCRIPTION:
The investigators will collect the blood samples at different time points: 0 hour, 2 hours, 4 hours, 6 hours, and 8 hours after the first time and the steady state concentration(more than 4 times drug administration) of drug administration from the patients receive treatment with CAZ-AVI to detect plasma drug concentrations of CAZ-AVI. The collected specimens will be stored in a refrigerator at 0-8 °C, centrifuges within 24 hours (4 °C, 4000 r/min, 10 min), and the supernatant will be collected in an EP tube and stored at -80°C until subsequent analysis. Ultra-high performance liquid chromatography-mass spectrometry (UPLC-MS/MS) will be used to detect plasma drug concentrations of CAZ-AVI. According to the outcomes ,the investigators will characterize the population pharmacokinetics (PPK) of CAZ-AVI in critically ill patients and performed pharmacodynamic target attainment analyses to determine optimal dosing regimens for patients with and without continuous renal replacement therapy (CRRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe sepsis and treated with ceftazidime avibactam
* Age ≥ 18 years
* The patient or authorized persons agree and sign the informed consent
* The patient's hemoglobin is greater than 70g/l during blood collection

Exclusion Criteria:

* The expected length of ICU stay less than 48 hours,
* Pregnant woman,
* The blood sample is hemolysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe sepsis and treatment with Ceftazidime-Avibactam in ICU of the First Affiliated Hospital of the Medical College of Zhejiang University from January 1, 2022 to September 30, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Plasma drug concentrations of CAZ-AVI | 0 hour, 2 hours, 4 hours, 6 hours, and 8 hours after the first time of drug administration
  Plasma drug concentrations of CAZ-AVI after the first time of drug administration
Plasma drug concentrations of CAZ-AVI | 0 hour, 2 hours, 4 hours, 6 hours, and 8 hours after the steady state concentration (more than 4 times drug administration) of drug administration
  Plasma drug concentrations of CAZ-AVI after the steady state concentration (more than 4 times drug administration) of drug administration
A population pharmacokinetic (PopPK) model for CAZ-AVI and to propose an appropriate dosing regimen in Chinese critically ill patients. | After obtaining the patient's plasma drug concentration
  By conducting pharmacokinetic and pharmacodynamic analysis on the plasma drug concentration data of patients receiving CAZ-AVI treatment in the intensive care unit, we aim to develop a population pharmacokinetic (PopPK) model for critically ill patients in China and to formulate an appropriate dosing regimen for critically ill patients with varying degrees of renal function, including those undergoing renal replacement therapy.

SECONDARY OUTCOMES:
Serum albumin | The day of the first time of drug administration
  The level of serum albumin on the day of the first time of drug administration
Serum albumin | The day of the steady state concentration (more than 4 times drug administration) of drug administration
  The level of serum albumin on the day of the steady state concentration(more than 4 times drug administration) of drug administration
The level of creatinine | The day of the first time of drug administration
  The level of creatinine on the day of the first time of drug administration
The level of creatinine | The day of the first time of the steady state concentration (more than 4 times drug administration) of drug administration
  The level of creatinine on the day of the steady state concentration(more than 4 times drug administration) of drug administration
The level of glomerular filtration rate | The day of the first time of drug administration
  The level of glomerular filtration rate on the day of the first time of drug administration
The level of glomerular filtration rate | The day of the steady state concentration (more than 4 times drug administration) of drug administration
  The level of glomerular filtration rate on the day of the steady state concentration (more than 4 times drug administration) of drug administration
Whether received renal replacement therapy | The day of the first time of drug administration
  Whether the patient received renal replacement therapy on the day of the first time of drug administration, and the results are recorded in the form of categorical variables,(e.g.,yes or no).
Whether received renal replacement therapy | The day of the steady state concentration (more than 4 times drug administration) of drug administration
  Whether the patient received renal replacement therapy on the day of the steady state concentration (more than 4 times drug administration) of drug administration, and the results are recorded in the form of categorical variables,(e.g.,yes or no).
Respiratory function | The day of the first time of administration
  Whether the patient received mechanical ventilation on the day of the first time of drug administration, and the results are recorded in the form of categorical variables,(e.g.,yes or no).
Respiratory function | The day of the steady state concentration (more than 4 times drug administration) of drug administration
  Whether the patient received mechanical ventilation on the day of the steady state concentration (more than 4 times drug administration) of drug administration, and the results are recorded in the form of categorical variables,(e.g.,yes or no).
Cardiovascular function | The day of the first time of drug administration
  Whether the patient received vasoactive agents(including norepinephrine, epinephrine, dobutamine, and metarylamine), and the results are recorded in the form of categorical variables,(e.g.,yes or no).
Cardiovascular function | The day of the steady state concentration (more than 4 times drug administration) of drug administration
  Whether the patient received vasoactive agents(including norepinephrine, epinephrine, dobutamine, and metarylamine), and the results are recorded in the form of categorical variables,(e.g.,yes or no).
CRRT treatment dosage | The day of the first time of drug administration
  The specific parameters for patients undergoing CRRT include the type of CRRT machine, treatment modality, treatment method, filter type, treatment duration, pre-dilution volume, post-dilution volume, blood pump flow rate, dialysis pump flow rate, average hourly fluid removal, treatment dose, ultrafiltration rate, and waste fluid volume
CRRT treatment dosage | The day of the steady state concentration (more than 4 times drug administration) of drug administration
  The specific parameters for patients undergoing CRRT include the type of CRRT machine, treatment modality, treatment method, filter type, treatment duration, pre-dilution volume, post-dilution volume, blood pump flow rate, dialysis pump flow rate, average hourly fluid removal, treatment dose, ultrafiltration rate, and waste fluid volume
microbiological clearance, infection-related mortality | 14 day after the onset of infection
  microbiological clearance, 14 day infection-related mortality,
all-cause mortality | 30 day and 90 day after the onset of infection
  30 day all-cause mortality,90 day all-cause mortality
length of stay | Day 1 is defined as the day of confirmed diagnosis, the duration from confirmed diagnosis to ICU discharge will be measured.
  Post-infection ICU length of stay
length of stay | From ICU admission to ICU discharge will be measured(assessed up to 120 days).
  Total ICU length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: YongHong Xiao, PhD, Study Chair — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital,College of Medicine,Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Respect ethics and protect patient privacy